CLINICAL TRIAL: NCT02554253
Title: The Impact of Ketamine on Postoperative Cognitive Dysfunction, Delirium, and Renal Dysfunction in Patients 75 Years of Age or Older and Undergoing Cardiac Surgery
Brief Title: The Impact of Ketamine on Postoperative Cognitive Dysfunction, Delirium, and Renal Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erica D. Wittwer, M.D., Ph.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-007148
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Results first posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Cognitive Disorders; Delirium; Acute Kidney Injury
MeSH Terms: conditions — Cognitive Dysfunction; Delirium; Acute Kidney Injury | interventions — Ketamine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ketamine (Active Comparator): Ketamine induction
  Interventions: Drug: Ketamine
- Propofol (Active Comparator): Propofol induction
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ketamine — Ketamine used for induction
  Other Names: Ketalar
  Arms: ketamine
Drug: Propofol — Propofol for induction
  Other Names: Diprivan; Propoven
  Arms: Propofol

SUMMARY:
Ketamine is a commonly used anesthetic medication which is used for induction of anesthesia as well as as an analgesic. It has been shown to have anti-inflammatory properties which may decrease post-operative complications following cardiac surgery with cardiopulmonary bypass that are thought to associated with inflammation. Some studies have shown that ketamine does decrease these complications when compared with anesthetics that are not commonly used in our cardiac anesthesiology practice. Propofol is another commonly used anesthetic medication which is used for induction of anesthesia. Ketamine has not been compared with propofol for potential to reduce post-operative complications associated with the inflammatory process. This study aims to see if ketamine will reduce the incidence of cognitive dysfunction, delirium, and renal dysfunction in comparison with propofol. In addition, the hemodynamic impact of ketamine compared propofol will be investigated.

ELIGIBILITY:
Scheduled to undergo cardiac surgery.

Inclusion criteria:

* age greater than or equal to 75 years presenting for cardiac surgery at the Mayo Clinic in Rochester, Minnesota;
* schedule to undergo complex cardiac surgery. Complex cardiac surgery will be defined as surgery involving more than one heart valve, redo-sternotomy procedures, or combined valvular and CABG procedures.

Exclusion criteria will include:

* left or right ventricular assist device implantation or explantation,
* procedures not requiring cardiopulmonary bypass,
* active infection or sepsis, severe hepatic disease or ascites,
* pre-operative renal dysfunction including a baseline creatinine equal to or greater than 1.5 mg/dL or requiring dialysis,
* immunosuppressive medication use (including steroid use),
* immunodeficiency syndrome,
* known neurologic or psychiatric disorder, or
* use of drugs for psychosis.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-09; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Wittwer, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were undergoing complex cardiac surgery at Mayo Clinic were recruited between August 2015 and October 2019.
Pre-assignment Details: Of the 265 patients assessed for eligibility, 52 were randomized to study groups. 8 did not meet inclusion criteria, 97 declined to participate, 96 were unable to be contacted before surgery, and 12 were unable to coordinate preoperative testing before surgery.
Period: Overall Study
Arm/Group | Ketamine | Propofol
Started | 26 | 26
Completed | 25 | 24
Not Completed | 1 | 2
Not completed — ineligible after enrollment | 1 | 0
Not completed — converted to transcatheter procedure | 0 | 1
Not completed — received both drugs | 0 | 1

BASELINE CHARACTERISTICS:
Population: 52 patients were enrolled. 3 patients did not complete the study. 1 patient was found to be ineligible after enrollment, 1 patient transitioned to a procedure that was in the exclusion criteria, and one patient received both the induction medications. This resulted in 25 patients for analysis in the ketamine group and 24 patients in the Propofol group.
Groups:
- Propofol: Propofol induction
  Propofol: Propofol used for induction
- Total: Total of all reporting groups
Arm/Group | Ketamine | Propofol | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.4 (3.5) | 76.1 (5.3) | 76.3 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 16 | 14 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 24 | 49
Trail Making Test A [Mean (Standard Deviation); unit: Z score] — Activity tests visual attention & task switching. Subjects connect 25 dots in numerical order as quickly and accurately as possible.
  Raw scores converted z-scores using published references. Z-score of zero corresponds to the mean score (time taken) in the reference population. Z-score of 1 indicates a value that is one standard deviation from the mean. A z-score greater than zero indicates a value above the mean (longer time, worse performance) and a score less than zero indicates a value below the mean (shorter time, better performance).
  1.5 or 2 SD from mean is usually considered impaired
  Z score | -0.1 (0.8) | 0 (1.1) | 0.0 (1.0)
Trail Making Test B [Mean (Standard Deviation); unit: Z score] — Activity tests visual attention & task switching. Subjects connect 25 dots in numerical order as quickly and accurately as possible.
  Raw scores converted z-scores using published references. Z-score of zero corresponds to the mean score (time taken) in the reference population. Z-score of 1 indicates a value that is one standard deviation from the mean. A z-score greater than zero indicates a value above the mean (longer time, worse performance) and a score less than zero indicates a value below the mean (shorter time, better performance).
  1.5 or 2 SD from mean is usually considered impaired
  Z score | 0.2 (1.0) | -0.1 (1.1) | 0.1 (1.1)
Hopkins Verbal Learning Test-Revised (HVLT-R) Learning Trials test [Mean (Standard Deviation); unit: Z score] — This activity tests the subject's ability to remember a list of 25 words read to the subject. This tests immediate recall of the words.
  Z-scores: the raw scores were converted z-scores using published references. Z-score of zero corresponds to the mean score (words recalled) in the reference population. Z-score of 1 indicates a value that is one standard deviation from the mean. A z-score greater than zero indicates a value above the mean (indicates better performance) and a score less than zero indicates a value below the mean (worse performance).
  Z score | -0.7 (0.9) | -0.5 (0.8) | -0.6 (0.9)
Hopkins Verbal Learning Test-Revised (HVLT-R) Delayed Recall [Mean (Standard Deviation); unit: Z score] — This activity tests the subject's ability to remember a list of 25 words 20-25 min after these words were previously read to the subject.
  Z-scores: the raw scores were converted z-scores using published references. Z-score of zero corresponds to the mean score (words recalled) in the reference population. Z-score of 1 indicates a value that is one standard deviation from the mean. A z-score greater than zero indicates a value above the mean (indicates better performance) and a score less than zero indicates a value below the mean (worse performance).
  Z score | -0.9 (1.3) | -0.8 (1.2) | -0.9 (1.2)
Hopkins Verbal Learning Test-Revised (HVLT-R) Digit Span [Mean (Standard Deviation); unit: Z score] — This activity tests the subject's ability to remember a list of numbers after the list is read to them. They are asked to repeat the numbers back in the same order presented.
  Z-scores: the raw scores were converted z-scores using published references. Z-score of zero corresponds to the mean score (words recalled) in the reference population. Z-score of 1 indicates a value that is one standard deviation from the mean. A z-score greater than zero indicates a value above the mean (indicates better performance) and a score less than zero indicates a value below the mean (worse performance).
  Z score | 0.2 (0.8) | 0.1 (1.0) | 0.2 (0.9)
Controlled Oral Word Association Test (COWAT) [Mean (Standard Deviation); unit: Z score] — This activity tests the subject's verbal fluency. They are given a category and asked to say as many words from that category as possible in a set timeframe.
  Z-scores: the raw scores were converted z-scores using published references. Z-score of zero corresponds to the mean score (words recalled) in the reference population. Z-score of 1 indicates a value that is one standard deviation from the mean. A z-score greater than zero indicates a value above the mean (indicates better performance) and a score less than zero indicates a value below the mean (worse performance).
  Z score | 0.1 (0.8) | 0.1 (0.8) | 0.1 (0.8)
Stroop color/word test [Mean (Standard Deviation); unit: Z score] — This tests the subject's ability to name the color a word is printed in when the word is the name of a different color. Example: Red printed in green ink, the answer is green.
  Z-scores: the raw scores were converted z-scores using published references. Z-score of zero corresponds to the mean score (words recalled) in the reference population. Z-score of 1 indicates a value that is one standard deviation from the mean. A z-score greater than zero indicates a value above the mean (indicates better performance) and a score less than zero indicates a value below the mean (worse performance).
  Z score | -0.3 (1.0) | -0.6 (1.3) | -0.4 (1.1)
Mini-Mental Status Exam [Mean (Standard Deviation); unit: Z score] — This 11 question exam tests multiple aspects of cognitive function including orientation, attention, memory, language, and visual spatial skills and only takes a few minutes.
  Z-scores: the raw scores were converted z-scores using published references. Z-score of zero corresponds to the mean score (words recalled) in the reference population. Z-score of 1 indicates a value that is one standard deviation from the mean. A z-score greater than zero indicates a value above the mean (indicates better performance) and a score less than zero indicates a value below the mean (worse performance).
  Z score | 0.7 (0.9) | 0.4 (1.1) | 0.6 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Postoperative Cognitive Dysfunction
Description: Pre and postoperative cognitive studies will be performed to assess change in cognitive function.
  Postoperative cognitive dysfunction (POCD) was defined a-priori as a decline of decline of >1 standard deviation (i.e. z-score decline of > 1) on at least 2 neurocognitive tests. The neurocognitive tests utilized include Trail making Test A, Trail making Test B, Hopkins Verbal Learning Test-Revised Learning trials, Hopkins Verbal Learning Test-Revised Delayed Recall, Digit Span, Controlled Oral Word Association Test, Stroop color/word test, and the Mini Mental Status Examination.
Time Frame: Baseline (preoperative cognitive tests) to hospital discharge or 10 days postoperatively whichever came first.
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Propofol
Number analyzed (Participants) | 25 | 24
Participants | 16 | 10
Statistical Analysis 1: Comparison: Ketamine vs Propofol; Raw scores converted to z-scores using published references. Percentage of patients experiencing a decline of > 1 standard deviation was compared between groups using Fisher's exact test. The outcome of postoperative cognitive dysfunction (POCD) was defined a-priori as a decline of decline of >1 standard deviation (i.e. z-score decline of > 1) on at least 2 neurocognitive tests and was compared between groups using Fisher's exact test; Test type: Superiority — Pilot study; p = 0.23, Fisher Exact

2. Secondary Outcome: Number of Patients With Acute Kidney Injury
Description: AKI was defined by Kidney Disease Improving Global Outcomes (KDIGO) criteria including an increase in serum creatinine ≥0.3 mg/dL within 48 hours, an increase in serum creatinine to ≥1.5 times baseline within 7 days, and urine output < 0.5 mL/kg/hr for 6 hours.
Time Frame: Baseline (preoperative cognitive tests) to hospital discharge or 10 days postoperatively whichever came first.
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Propofol
Number analyzed (Participants) | 25 | 24
Participants | 6 | 12
Statistical Analysis 1: Comparison: Ketamine vs Propofol; Test type: Superiority; p = 0.08, Fisher Exact

3. Secondary Outcome: Number of Patients Who Develop Postoperative Delirium
Description: Delirium was defined as a positive CAM (Confusion assessment method) score. CAM score was recorded every 12 hours postoperatively as per routine. The CAM consists of 4 features: 1-Onset, 2-Inattention, 3-Disorganized thinking, and 4-altered level of consciousness. The diagnosis of delirium by CAM is based on the presence of features 1 and 2, and either 3 or 4. The score is either positive or negative. Positive means the patient has delirium and negative indicates the patient is not delirious.
Time Frame: Baseline (preoperative cognitive tests) to hospital discharge or 10 days postoperatively whichever came first.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Propofol
Number analyzed (Participants) | 25 | 24
Participants | 0 | 1
Statistical Analysis 1: Comparison: Ketamine vs Propofol; Test type: Superiority; p = 0.31, Chi-squared

ADVERSE EVENTS:
Time Frame: Surgery to discharge, up to 10 days postoperatively
Arm/Group | Ketamine | Propofol
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=25) | Propofol (N=24)
Complete heart block (Cardiac disorders) | 0 (0) | 1 (1)
RV failure (Cardiac disorders) | 1 (1) | 0 (0) — Post bypass right ventricular failure requiring IABP
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Respiratory failure one week post op requiring reintubation
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Ileus and intestinal perforation requiring surgery
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Not powered to detect differences in acute kidney injury. A larger study will be needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT02554253/Prot_SAP_000.pdf